CLINICAL TRIAL: NCT03456102
Title: Statin Adjunctive Therapy for TB (StAT- TB)
Brief Title: Statin Adjunctive Therapy for TB
Acronym: StAT-TB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00145353
Record Dates: First submitted 2018-02-19; First posted 2018-03-07 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pravastatin 80 mg (Other): Pravastatin 80 mg, isoniazid 300 mg, rifampin 450 mg (weight <50 kg) or 600 mg (weight >50 kg), pyrazinamide 20-25 mg/kg, and ethambutol 15-20 mg/kg daily for 14 days Arm 2 will only be recruited if pravastatin 40 mg is well tolerated and safe, yet drug exposures are significantly reduced due to the known interaction with rifampin.
  Interventions: Drug: Pravastatin
- Pravastatin 120 mg (Other): Pravastatin 120 mg, isoniazid 300 mg, rifampin 450 mg (weight <50 kg) or 600 mg (weight >50 kg), pyrazinamide 20-25 mg/kg, and ethambutol 15-20 mg/kg daily for 14 days Arm 3 will only be recruited if pravastatin 80 mg is well tolerated and safe, yet drug exposures are significantly reduced due to the known interaction with rifampin.
  Interventions: Drug: Pravastatin
- Pravastatin 160 mg (Other): Pravastatin 160 mg, isoniazid 300 mg, rifampin 450 mg (weight <50 kg) or 600 mg (weight >50 kg), pyrazinamide 20-25 mg/kg, and ethambutol 15-20 mg/kg daily for 14 days Arm 4 will only be recruited if pravastatin 120 mg is well tolerated and safe, yet drug exposures are significantly reduced due to the known interaction with rifampin.
  Interventions: Drug: Pravastatin
- Pravastatin 40 mg (Other): Pravastatin 40 mg, isoniazid 300 mg, rifampin 450 mg (weight <50 kg) or 600 mg (weight >50 kg), pyrazinamide 20-25 mg/kg, and ethambutol 15-20 mg/kg daily for 14 days
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Pravastatin — Phase IIB clinical trial: A two-week safety/PK study to determine pravastatin exposures over 24 hours when given together with first-line treatment (HRZE) and ensure the combination is safe and well-tolerated.
  A two-week safety/PK study to determine pravastatin exposures over 24 hours when given together with first-line treatment (HRZE) and ensure the combination is safe and well-tolerated.

SUMMARY:
There is an urgent need for novel therapies to shorten TB treatment and improve long-term lung function outcomes. Host-directed therapies (HDT) have received significant attention recently given the ability of M. tuberculosis to subvert host immune responses and cause destructive lung pathology. Statins are among the most promising HDT agents for TB. In addition to having a highly favorable safety profile, statins have been shown to have anti-TB activity in macrophages, to synergize with anti-TB drugs, and to shorten the duration of TB treatment in the standard mouse model.

The StAT-TB trial will comprise two different stages. In the 14-day Stage 1 study, investigators will test the safety and tolerability, as well as Pharmacokinetics (PK), of two different doses of pravastatin co-administered with standard anti-TB treatment. In Stage 2, investigators will test the ability of pravastatin adjunctive therapy (dose to be determined in Stage 1) to shorten the mean time to sputum culture conversion (primary endpoint) and improve lung function outcomes (secondary endpoints) relative to the standard regimen. In addition, investigators will continue to investigate the anti-TB mechanism of action of pravastatin in order to further improve HDT options for TB in the future.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Clinical signs and symptoms of pulmonary tuberculosis
* Abnormal chest radiograph consistent with pulmonary tuberculosis
* At least one sputum positive for M. tuberculosis by Xpert Mycobacterium tuberculosis (MTB)/resistance to rifampicin (RIF) with a cycle threshold (Ct) <28.
* Documentation of HIV status
* Weight ≥45 kg
* Karnofsky score of at least 60
* Ability to provide informed consent
* Ability to adhere to study follow-up visits
* Ability to adhere to contraceptive requirements and willing to use two forms of contraception.
* Five days or fewer of anti-tuberculosis treatment within the previous 3 months

Exclusion Criteria:

* A history of severe adverse reactions to any statin or any other study agent or contraindications to use of statins.
* Current use of statins or other lipid-lower agents;
* Clinical indication for statin therapy based on cardiovascular risk (Familial hypercholesterolemia, Previous history of myocardial infarction or stroke)
* For HIV-positive individuals, a cluster of differentiation 4 (CD4+) T-cell count <100/mm3
* Use of antiretroviral drugs
* Hemoglobin concentration less than 7 g/dL;
* Baseline creatinine kinase elevation more than three times the upper limit of normal
* Abnormal baseline laboratory values (Baseline alanine aminotransferase (ALT) concentration more than three times the upper limit of normal, Serum creatinine concentration more than twice the upper limit of normal, Serum total bilirubin level greater than twice the upper limit of normal, Platelet count < 100,000/mm3, White Blood Cell (WBC) < 2500 (mcL))
* Pregnant or breastfeeding;
* Silico-tuberculosis.
* Currently receiving TB treatment
* Concomitant disorders or conditions for which isoniazid, rifampin, pyrazinamide, or ethambutol is contraindicated. These include sever hepatic damage, acute liver disease of any cause, acute uncontrolled gouty arthritis and peripheral neuropathy.
* Any medical or psychological condition which, in the view of the study investigator, makes study participation inadvisable.
* Infection with an isolate known to be resistant to a first -line TB drug; for example rifampin.
* More than five days of anti-tuberculosis treatment within the previous 3 months
* Planned or current use of cyclosporine, tacrolimus, erythromycin or colchicine
* Central nervous system (CNS) TB
* Extra-pulmonary TB only, not in combination with pulmonary TB
* History of TB

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Chaisson, Principal Investigator — Johns Hopkins University
Locations (1):
- Chris Hani Baragwanath Hospital, Johannesburg, South Africa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from clinics in Soweto, South Africa by the study team at the PHRU, Chris Hani Baragwanath Academic Hospital, Soweto, South Africa. Participants were recruited based on having a sputum specimen that is positive for TB by GeneXpert MTB/RIF.
Groups:
- Pravastatin 40 mg: Pravastatin 40 mg, isoniazid 300 mg, rifampin 450 mg (weight <50 kg) or 600 mg (weight >50 kg), pyrazinamide 20-25 mg/kg, and ethambutol 15-20 mg/kg daily for 14 days Arm 4 will only be recruited if pravastatin 80 mg is not tolerated as specified in protocol.
  Pravastatin: Phase IIB clinical trial: A two-week safety/PK study to determine pravastatin exposures over 24 hours when given together with first-line treatment (HRZE) and ensure the combination is safe and well-tolerated.
  A two-week safety/PK study to determine pravastatin exposures over 24 hours when given together with first-line treatment (HRZE) and ensure the combination is safe and well-tolerated.
- Pravastatin 80 mg: Pravastatin 80 mg, isoniazid 300 mg, rifampin 450 mg (weight <50 kg) or 600 mg (weight >50 kg), pyrazinamide 20-25 mg/kg, and ethambutol 15-20 mg/kg daily for 14 days Arm 2 will only be recruited if pravastatin 80 mg is well tolerated and safe, yet drug exposures are significantly reduced due to the known interaction with rifampin.
  Pravastatin: Phase IIB clinical trial: A two-week safety/PK study to determine pravastatin exposures over 24 hours when given together with first-line treatment (HRZE) and ensure the combination is safe and well-tolerated.
  A two-week safety/PK study to determine pravastatin exposures over 24 hours when given together with first-line treatment (HRZE) and ensure the combination is safe and well-tolerated.
- Pravastatin 120 mg: Pravastatin 120 mg, isoniazid 300 mg, rifampin 450 mg (weight <50 kg) or 600 mg (weight >50 kg), pyrazinamide 20-25 mg/kg, and ethambutol 15-20 mg/kg daily for 14 days Arm 3 will only be recruited if pravastatin 120 mg is well tolerated and safe, yet drug exposures are significantly reduced due to the known interaction with rifampin.
  Pravastatin: Phase IIB clinical trial: A two-week safety/PK study to determine pravastatin exposures over 24 hours when given together with first-line treatment (HRZE) and ensure the combination is safe and well-tolerated.
  A two-week safety/PK study to determine pravastatin exposures over 24 hours when given together with first-line treatment (HRZE) and ensure the combination is safe and well-tolerated.
- Pravastatin 160 mg: Pravastatin 160 mg, isoniazid 300 mg, rifampin 450 mg (weight <50 kg) or 600 mg (weight >50 kg), pyrazinamide 20-25 mg/kg, and ethambutol 15-20 mg/kg daily for 14 days
  Pravastatin: Phase IIB clinical trial: A two-week safety/PK study to determine pravastatin exposures over 24 hours when given together with first-line treatment (HRZE) and ensure the combination is safe and well-tolerated.
  A two-week safety/PK study to determine pravastatin exposures over 24 hours when given together with first-line treatment (HRZE) and ensure the combination is safe and well-tolerated.
Period: Overall Study
Arm/Group | Pravastatin 40 mg | Pravastatin 80 mg | Pravastatin 120 mg | Pravastatin 160 mg
Started | 10 | 6 | 0 | 0
Completed | 10 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled and no data was collected in the 120mg and 160mg pravastatin arms due to early termination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pravastatin 40 mg | Pravastatin 80 mg | Pravastatin 120 mg | Pravastatin 160 mg | Total
Number analyzed (Participants) | 10 | 6 | 0 | 0 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.70 (5.35) | 26.83 (7.03) |  |  | 26.75 (5.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 |  |  | 5
  Male | 7 | 4 |  |  | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African/Black | 10 | 6 |  |  | 16
  Coloured | 0 | 0 |  |  | 0
  Indian/Asian | 0 | 0 |  |  | 0
  White | 0 | 0 |  |  | 0
  Other | 0 | 0 |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 10 | 6 |  |  | 16
Weight at Baseline (kg) [Count of Participants; unit: Participants]
  45-49kg | 1 | 0 |  |  | 1
  50-59kg | 7 | 4 |  |  | 11
  60-69kg | 2 | 2 |  |  | 4
HIV Status [Count of Participants; unit: Participants]
  Negative | 10 | 6 |  |  | 16
  Positive | 0 | 0 |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety of Escalating Doses of Pravastatin as Assessed by Number of Adverse Events
Description: Safety of escalating doses of pravastatin (40 mg - 160 mg) when co-administered with rifampin, as evidenced by number of Grade 3 or higher adverse events.
Time Frame: Up to 30 days
Population: Participants were not enrolled in Arms 3 and 4 due to early termination.
Measure: Number; unit: AEs Grade 3 or Higher
Groups:
- Pravastatin 40 mg: Pravastatin 40 mg, isoniazid 300 mg, rifampin 450 mg (weight <50 kg) or 600 mg (weight >50 kg), pyrazinamide 20-25 mg/kg, and ethambutol 15-20 mg/kg daily for 14 days
  Pravastatin: Phase IIB clinical trial: A two-week safety/PK study to determine pravastatin exposures over 24 hours when given together with first-line treatment (HRZE) and ensure the combination is safe and well-tolerated.
  A two-week safety/PK study to determine pravastatin exposures over 24 hours when given together with first-line treatment (HRZE) and ensure the combination is safe and well-tolerated.
- Pravastatin 80 mg: Pravastatin 80 mg, isoniazid 300 mg, rifampin 450 mg (weight <50 kg) or 600 mg (weight >50 kg), pyrazinamide 20-25 mg/kg, and ethambutol 15-20 mg/kg daily for 14 days Arm 2 will only be recruited if pravastatin 40 mg is well tolerated and safe, yet drug exposures are significantly reduced due to the known interaction with rifampin.
  Pravastatin: Phase IIB clinical trial: A two-week safety/PK study to determine pravastatin exposures over 24 hours when given together with first-line treatment (HRZE) and ensure the combination is safe and well-tolerated.
  A two-week safety/PK study to determine pravastatin exposures over 24 hours when given together with first-line treatment (HRZE) and ensure the combination is safe and well-tolerated.
- Pravastatin 120 mg: Pravastatin 120 mg, isoniazid 300 mg, rifampin 450 mg (weight <50 kg) or 600 mg (weight >50 kg), pyrazinamide 20-25 mg/kg, and ethambutol 15-20 mg/kg daily for 14 days Arm 3 will only be recruited if pravastatin 80 mg is well tolerated and safe, yet drug exposures are significantly reduced due to the known interaction with rifampin.
  Pravastatin: Phase IIB clinical trial: A two-week safety/PK study to determine pravastatin exposures over 24 hours when given together with first-line treatment (HRZE) and ensure the combination is safe and well-tolerated.
  A two-week safety/PK study to determine pravastatin exposures over 24 hours when given together with first-line treatment (HRZE) and ensure the combination is safe and well-tolerated.
- Pravastatin 160 mg: Pravastatin 160 mg, isoniazid 300 mg, rifampin 450 mg (weight <50 kg) or 600 mg (weight >50 kg), pyrazinamide 20-25 mg/kg, and ethambutol 15-20 mg/kg daily for 14 days Arm 4 will only be recruited if pravastatin 120 mg is well tolerated and safe, yet drug exposures are significantly reduced due to the known interaction with rifampin.
  Pravastatin: Phase IIB clinical trial: A two-week safety/PK study to determine pravastatin exposures over 24 hours when given together with first-line treatment (HRZE) and ensure the combination is safe and well-tolerated.
  A two-week safety/PK study to determine pravastatin exposures over 24 hours when given together with first-line treatment (HRZE) and ensure the combination is safe and well-tolerated.
Arm/Group | Pravastatin 40 mg | Pravastatin 80 mg | Pravastatin 120 mg | Pravastatin 160 mg
Number analyzed (Participants) | 10 | 6 | 0 | 0
AEs Grade 3 or Higher | 8 | 4 |  |

ADVERSE EVENTS:
Time Frame: Up to 5 months.
Description: No patients were enrolled in Study Arms 3 and 4 due to early termination.
Arm/Group | Pravastatin 40 mg | Pravastatin 80 mg | Pravastatin 120 mg | Pravastatin 160 mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 4/10 | 1/6 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 5/10 | 3/6 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pravastatin 40 mg (N=10) | Pravastatin 80 mg (N=6) | Pravastatin 120 mg (N=0) | Pravastatin 160 mg (N=0)
Elevated Uric Acid (Investigations) | 3 (3) | 1 (1) | NA | NA
Elevated liver enzymes (ALT/AST) (Investigations) | 1 (1) | 0 (0) | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pravastatin 40 mg (N=10) | Pravastatin 80 mg (N=6) | Pravastatin 120 mg (N=0) | Pravastatin 160 mg (N=0)
Elevated liver enzymes (ALT/AST) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated creatinine kinase (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated uric acid (Investigations) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Decreased hemoglobin level (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT03456102/Prot_SAP_000.pdf